CLINICAL TRIAL: NCT06924008
Title: Development of an Intervention Aimed at Facilitating the Use of Eye Contact in Adults With Autism: A Qualitative Study With Methodological Triangulation
Brief Title: Developing an Intervention Facilitating the Use of Eye Contact in Adults With Autism
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Dimence Groep (Unknown)
Responsible Party: Principal Investigator, Jos Boer, MSc, UMC Utrecht
Other Study IDs: 559903; Dimence Groep (Other: Dimence Groep)
Record Dates: First submitted 2025-03-28; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder (ASD); Relative (Related Person); Care Giver
Keywords: Intervention; Eye contact; Autism Spectrum Disorder; ASD; Intervention Mapping
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to develop a methodological intervention for adults with autism that will help them reduce problems arising from eye contact.

DETAILED DESCRIPTION:
Eye contact is fundamental to human interaction, not only in terms of the experience of connection with others, but also in terms of cognitive skills and social-emotional development. In adults with autism, eye contact is sometimes atypical, which in individual cases can lead to problems in the aforementioned areas. An intervention could possibly lead to a reduction of these problems. However, to date, there is no insight into the problems that this population experiences due to eye contact, how this differs from people without autism, to what extent adults with autism wish to optimize eye contact with others, what they themselves see as solutions for this, and when it proves fruitful to develop an intervention based on all these facets; what an effective intervention could be for this (and who the target group is). While insight into all of this could lead to a reduction in problems that adults with autism and/or their interaction partner experience due to their eye contact. To gain this insight, it is necessary to inventory, among both adults with and without autism, what problems adults with autism actually experience with regard to eye contact, and what their ideas are to reduce these problems. In addition, it is necessary to investigate in a substantiated methodical way which intervention forms a solution for the distilled problems and to test these, in order to be able to assess their effectiveness. If effective, then this intervention could at least contribute to the well-being of adults with autism and a mutually pleasant contact with interaction partners. The current study aims to provide for this and to arrive at an effective intervention that will help adults with autism experience less difficulty as a result of eye contact.

The research design chosen is qualitative research using triangulation by means of descriptive research in the form of semi-structured interviews and Intervention Mapping. The interviews have now taken place. These interviews, in addition to available scientific literature on eye contact in adults with autism, form the starting point for intervention development by means of Intervention Mapping. Intervention Mapping was chosen because the goal is to develop an intervention that will later be as effective as possible. This can be achieved by carefully weighing and substantiating the choices for the goal and the approach in the design phase. Intervention Mapping provides a theoretical basis for the intervention, which makes it more likely that the intervention will also work in practice. In addition, it provides a systematically described intervention and an implementation plan, making the intervention transferable and easier to put into practice. A major advantage of Intervention Mapping is that attention is paid to the way in which the results and effects of the project should be evaluated later, already in the development phase. In this way, Intervention Mapping contributes to increasing the effectiveness of the project. The aim of Intervention Mapping is to provide a framework for effective decision-making at every step of planning, implementation and evaluation. The Intervention Mapping protocol consists of six steps, with a number of tasks described for each step. Although Intervention Mapping is presented as a series of steps, it can be seen as iterative rather than linear. Programme planners switch back and forth between tasks and steps. The process is also cumulative: each step is based on previous steps.

ELIGIBILITY:
Inclusion criteria for adults with autism

* Adults classified with autism, determined according to an internationally recognized classification system.
* Outpatient treatment within a specialized autism center in the Netherlands.
* Able to understand the topics to be discussed.
* Motivation to participate in research.

Exclusion criteria for adults with autism

* No good command of the Dutch language.
* Use of alcohol and/or recreational drugs during the study.
* Mentally too unstable to participate in the study.
* Familiarity with treatment in the VGZ.

Inclusion criteria for those involved

* Adults without DSM classification.
* Living in the Netherlands.
* Able to understand the topics to be discussed.
* Motivation to participate in research.

Exclusion criteria for those involved

* No good command of the Dutch language.
* Use of alcohol and/or recreational drugs during the study.

Inclusion criteria for healthcare providers

* Practicing psychiatrist, clinical psychologist or nurse specialist at an autism expertise center in the Netherlands.
* Living in the Netherlands.
* Motivation to participate in research.

Exclusion criteria for healthcare providers

- No good command of the Dutch language.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults with autism, caregivers of adults with autism, and healthcare providers (psychiatrists, psychologists and nursing specialists in psychiatry).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2026-07-03 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Developing an intervention using the Intervention Mapping method. | Up to 12 months.
  An effective intervention for adults with autism that reduces their difficulty with eye contact problems, with use of Intervention Mapping.
  The Intervention Mapping protocol consists of six steps, with a number of tasks described for each step. These steps are carried out within focus groups, with two months of time set aside for each step.
  The six steps of the Intervention Mapping process are:
  Step 1: Needs assessment Step 2: Change objectives Step 3: Theoretical methods and practical techniques Step 4: Programme design and production Step 5: Program Adoption and Implementation Step 6: Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Nynke Boonstra, Professor, Study Chair — UMC Utrecht
Locations (1):
- Dimence Groep, Deventer, Overijssel, Netherlands